## Title of the study

## Efficacy of atorvastatin versus colchicine in reducing myocardial damage biomarkers in patients with rheumatoid arthritis, with severe activity, pilot study.

Name of the Document

**Statistical Analysis Plan** 

Date of the document

July 25, 2018

## STATISTIC ANALYSIS.

The variables will be described by means of frequencies or percentages. The statistical analysis of each variable will be carried out with measures of central tendency and dispersion, the normality of the data will be evaluated. The variables with normal distribution will be expressed as mean and standard deviation. The qualitative data will be expressed as a percentage and frequency distribution. T student analysis of the means will be performed. A p less than 0.05 will be taken as statistical significance. All this will be done through the statistical program R version 3.4.3.

## SAMPLE'S SIZE CALCULATION

Initially, a pilot study with 30 patients per group, according to Browne, will be recalculated based on the preliminary result and the power of the effect.